CLINICAL TRIAL: NCT01047800
Title: Effectiveness of Counseling for Functional Gastrointestinal Disorder Patients: A Double-blind Randomized Controlled Trial
Brief Title: Functional Gastrointestinal Disorder Screening Program - A Randomized Controlled Trial
Acronym: FGISP-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Justin Che-Yuen Wu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: FGISP-RCT
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Non-erosive Gastroesophageal Reflux Disease; Functional Dyspepsia; Irritable Bowel Syndrome
Keywords: Functional gastrointestinal disorder; GERD; reflux; irritable bowel syndrome; Functional dyspepsia; postprandial fullness; counseling; service
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases; Gastroesophageal Reflux | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling group (Experimental): Two extra counseling sessions will be arranged for the Counseling group immediately after visiting the physician
  Interventions: Behavioral: Counseling
- Control (No Intervention): Usual management in GI specialty clinic

INTERVENTIONS:
Behavioral: Counseling — Two extra counseling sessions will be arranged for the Counseling group immediately after visiting the physician in First and Final visits. Each session lasts for about 15 minutes with the following content:
  First visit: prevalence of FGID in Hong Kong, chronicity nature of the disease, negative endoscopy result to be expected, time to answer patient's questions
  Final visit : prevalence of FGID in Hong Kong (reinforcement), chronicity nature of the disease (reinforcement), explanation of the endoscopy result, management of disease via lifestyle modification, use of medication, need for further or repeated investigation, time to answer patient's questions.
  Arms: Counseling group

SUMMARY:
Background:

Functional gastrointestinal disorder (FGID) is the most common gastrointestinal disease in daily clinical practice. The disease is symptomatic but has no identifiable cause by standard diagnostic tests such as endoscopy. It is characterized by its frequent relapses and thus the disease causes a significant level of stress and anxiety to patients. Due to the complexity and chronicity of the disease, it is believed that appropriate counseling on the nature and management of the disease is necessary to decrease patient's anxiety level and improve quality of life.

Indication:

Patients who have symptoms suggestive of FGID including non-erosive gastroesophageal reflux disease (NERD), functional dyspepsia (FD) or irritable bowel syndrome (IBS).

Aim:

To validate the effectiveness of counseling in patients suffering from FGID.

Method:

Patients recruited to the study will follow the usual management of patients attending the Gastroenterology specialty clinic in Prince of Wales Hospital. Standard blood tests and endoscopy will be performed. Standard medication will be given to the patients for 8 weeks after endoscopy and the patients will come back to the specialty clinic for a final visit.

The patient will be given an "on-demand follow up within 1 year" option at final visit. The patient will decide if he/she wants to come back to our specialty clinic to follow up his/her problem within one year.

Follow-up after Final Visit Follow-up questionnaires will be mailed to patients 6 months, 1 and 2 years after Final visit.

Randomization:

All the patients will be randomized into two groups in First Visit: 1) Control group, and 2) Counseling group. Both groups of patients will follow the above protocol, except that 2 extra counseling sessions will be arranged for the Counseling group immediately after visiting the physician.

DETAILED DESCRIPTION:
Patients recruited to the study will follow the usual management of patients attending the Gastroenterology specialty clinic in Prince of Wales Hospital, along with the following protocol:

First Visit

* Patient signs written consent
* Attending physician manages patient as usual
* Blood tests will be arranged for patient:

  * FD & NERD patients: CBC w/ differential count, LFT, TFT, random glucose
  * IBS patients: CBC w/ differential count, LFT, TFT, ESR, C-reactive protein
* Patient completes questionnaires

Endoscopy Visit

* Endoscopy examinations

  * FD & NERD patients: oesophagogastroduodenoscopy (OGD) with rapid urea test (RUT) and biopsy of antrum sample for histology to check h. pylori status
  * IBS patients: colonoscopy
* If no organic causes are found to explain for FGI symptoms, the following standard medication will be prescribed for 8 weeks:

FD: Pantoprazole 40mg daily; GERD: Pantoprazole 40mg daily; IBS: Mebeverine 135mg tid PRN before meal, Loperamide 4mg tid PRN (for diarrhea), Metamucil 2 teaspoon bid (for constipation).

Final Visit (8 weeks after endoscopy visit)

* Attending physician manages patient as usual
* Printout of investigation (endoscopy, blood tests) reports given to patient
* Patient completes questionnaires

The patient will be given an "on-demand follow up within 1 year" option at this visit. The patient will decide if he/she wants to come back to our specialty clinic to follow up his/her problem within one year. If the patient does not come back during this period, his/her case will be closed and a new referral will be required if he/she wants to be taken care by the specialty again.

Follow-up after Final Visit:

Follow-up questionnaires will be mailed to patients 6 months, 1 and 2 years after Final visit.

Randomization:

All the patients will be randomized into two groups in First Visit: 1) Control group, and 2) Counseling group. Both groups of patients will follow the above protocol, except that 2 extra counseling sessions will be arranged for the Counseling group immediately after visiting the physician:

Counseling at first visit:

- Contents include: prevalence of FGID in Hong Kong, chronicity nature of the disease, negative endoscopy result to be expected, time to answer patient's questions

Counseling at final visit:

- Contents include: prevalence of FGID in Hong Kong (reinforcement), chronicity nature of the disease (reinforcement), explanation of the endoscopy result, management of disease via lifestyle modification, use of medication, need for further or repeated investigation, time to answer patient's questions.

A research personnel who has been working with patients with FGID for at least one year will be responsible for the counseling service.

The random allocation sequence will be obtained from a computer-generated list of random numbers in blocks of 10 supplied by a trial statistician. Concealed allocation is achieved by an independent research staff who assigns intervention group according to consecutive numbers in sealed envelopes. The patients will be invited to participate in the study to assess 1 of 2 potentially helpful interventions. They will be explained that the relative effectiveness of both interventions are unproven and may or may not be beneficial.

In this study, the patients, attending physicians and endoscopes will all be blinded to the randomized arm that the patients are assigned to. The nature of the two arms will also be blinded to them. This arrangement is essential in clinical trials comparing different services or managing strategies and is clearly specified in the Patient Information Sheet.

ELIGIBILITY:
Inclusion Criteria:

Present with symptoms suggestive of any of the following FGID according to Rome III Classification:

* Non-erosive gastroesophageal reflux disease (NERD) Weekly symptoms of heartburn or acid regurgitation of moderate severity for at least 6 months
* Functional dyspepsia (FD) Weekly symptoms of epigastric burning sensation, early satiety or postprandial fullness for at least 6 months
* Irritable bowel syndrome (IBS)

Symptoms of abdominal pain or discomfort of at least 3 times a month, in the last 6 months, associated with 2 or more of the following:

* Improvement with defecation
* Onset associated with a change in frequency of stool
* Onset associated with a change in form (appearance) of stool

Exclusion Criteria:

* Erosive esophagitis (Still eligible for IBS patients)
* Peptic ulcer (Still eligible for IBS patients after complete ulcer healing)
* H. pylori positive
* Organic causes of symptoms, including malignancy, abnormal thyroid function, and inflammatory bowel disease.
* Previous gastric surgery
* Pregnancy
* Illiterate
* Unable to sign the written consent form • Abdominal surgery within one year prior to joining the program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Self-efficacy and decrease in psychological distress measured by Health status and management scales and Patient Health Questionnaire (PHQ) | 6 months after Final visit
Rate of attendance to "on-demand follow up within 1 year" option given at Final visit | 1 year after Final visit

SECONDARY OUTCOMES:
Frequency of doctor's visits | 1 and 2 years after Final visit
Use of emergency service | 1 and 2 years after Final visit
Self-rated health measured by Health status and management scales | 6 months, 1 and 2 years after Final visit
Social/role activities limitation measured by Health status and management scales | 6months, 1 and 2 years after Final visit

CONTACTS AND LOCATIONS:
Overall Officials: Justin C.Y. Wu, MBChB(CUHK), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No